CLINICAL TRIAL: NCT03435315
Title: Treadmill Exercise in Metabolic Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped prior to enrolling anticipated sample size due to COVID-19
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018P000014
Record Dates: First submitted 2018-01-23; First posted 2018-02-19 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill exercise (Active Comparator)
  Interventions: Other: Treadmill Exercise- traditional approach
- Treadmill exercise with behavioral techniques (Experimental)
  Interventions: Other: Treadmill Exercise- behavioral approach

INTERVENTIONS:
Other: Treadmill Exercise- behavioral approach — 12-session, 6-week treadmill exercise program utilizing behavioral techniques while walking
  Arms: Treadmill exercise with behavioral techniques
Other: Treadmill Exercise- traditional approach — 12-session, 6-week traditional treadmill exercise program
  Arms: Treadmill exercise

SUMMARY:
The main purpose of this study is to better understand the effects of two types of treadmill exercise programs that include education and/or techniques that may be helpful for exercise among individuals with, or at risk for, metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Referred by healthcare provider and given medical clearance for moderate-intensity exercise
2. Metabolic syndrome, defined as meeting three or more of the following criteria:

   * Obesity or overweight defined as BMI > 25
   * Impaired glycemia (fasting blood sugar of ≥ 100 [5.6 mmol/L] or glycated hemoglobin [A1C] of ≥ 5.7)
   * Increased blood pressure (130/85 mmHg or higher) or if you take medicine for high blood pressure
   * Increased fasting levels of triglycerides (≥ 150 or 1.7 mmol/L) or decreased fasting high-density lipoprotein (HDL) cholesterol (less than 40 mg/dL or 1 mmol/L for men or 50 mg/dL or 1.3 mmol/L for women) or if you take any medicines for dyslipidemia
3. Between the ages of 18-65
4. No regular physical activity (≥ 3 or more days per week) for the past 3 months

Exclusion Criteria:

1. Contraindications for treadmill exercise determined by their physician (e.g., cardiopulmonary limitations or diagnoses) or other inability to do treadmill exercise (e.g., musculoskeletal restrictions or severe balance impairment)
2. Confirmed diagnosis of coronary artery disease
3. Confirmed diagnosis of diabetes
4. Currently taking a beta blocker or calcium channel blocker medication
5. Uncontrolled and untreated hypertension, defined as a resting blood pressure of 150/90
6. Confirmed diagnosis of chronic obstructive pulmonary disease or other severe lung dysfunction that may interfere with exercise (e.g., severe asthma)
7. Self-reported psychotic disorder
8. Current practice of mindfulness mediation or mindful movement (e.g., yoga or tai chi), defined as regular daily practice or >2 classes or self-guided sessions per week in the past three months.
9. Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Recruitment Feasibility | Through study completion, an average of 1 year
  % willing to be randomized
Protocol Adherence | Through study completion, an average of 1 year
  % sessions attended

SECONDARY OUTCOMES:
Cardiopulmonary Dynamics | Weeks 1 and 6
  CardioPulmonary Exercise Testing (standard metabolic cart)
Fatigue | Week 0, week 3, post-intervention (after 6 week intervention)
  Fatigue Severity Scale-7; total score range: 7-49, higher scores = greater fatigue severity
Global Health | Week 0, week 3, post-intervention (after 6 week intervention)
  PROMIS Global Health-10; Global physical health total score range: 4-20, higher scores = better global physical health
Psychological Symptoms | Week 0, week 3, post-intervention (after 6 week intervention)
  Depression Anxiety and Stress Scale-21; Depression total score range: 0-21, higher scores = greater depressive symptoms
Affect | Week 0, week 3, post-intervention (after 6 week intervention)
  Positive and Negative Affect Schedule; 2 subscales; each with score range 10-50, higher = greater positive or negative affect
Anxiety Sensitivity | Week 0, week 3, post-intervention (after 6 week intervention)
  Anxiety Sensitivity Index-3; Total score range: 0-72, higher scores = higher levels of anxiety sensitivity
Distress Tolerance | Week 0, week 3, post-intervention (after 6 week intervention)
  Distress Tolerance Scale; total score range: 15-75, higher scores = higher levels of distress tolerance
Discomfort Intolerance | Week 0, week 3, post-intervention (after 6 week intervention)
  Discomfort Intolerance Scale-Revised; total score range: 0-126, higher scores = higher levels of discomfort intolerance
Physical Activity Acceptance | Week 0, week 3, post-intervention (after 6 week intervention)
  Physical Activity Acceptance Questionnaire; total score range: 10-70, higher scores = greater physical activity acceptance
Exercise Self-Efficacy | Week 0, week 3, post-intervention (after 6 week intervention)
  Multidimensional Self-Efficacy Scale; total score range: 0-90, higher scores = higher levels of exercise self-efficacy
Exercise Motivation | Week 0, week 3, post-intervention (after 6 week intervention)
  Behavioral Regulation towards Exercise Questionnaire-2; 5 subscales, each with score range: 0-16, higher scores = higher levels of regulation
Exercise Barriers | Week 0, week 3, post-intervention (after 6 week intervention)
  Exercise Benefits and Barriers Scale; 2 subscales; Exercise benefits subscale score range: 29-116, higher scores = higher perceived benefit from exercise; Exercise barriers subscale score range: 14-56, higher scores = higher perceived barriers to exercise
Physical Activity | Week 0, week 3, post-intervention (after 6 week intervention)
  Godin Leisure Time Exercise Questionnaire; open-ended responses, higher scores = greater activity time
Trait Mindfulness | Week 0, week 3, post-intervention (after 6 week intervention)
  Five Facet Mindfulness Questionnaire; 5 subscales; Observe subscale score range: 8-40, higher scores = greater observing skills; Describe subscale score range: 8-40, higher scores = greater describing skills; Acting with Awareness subscale score range: 8-40, higher scores = greater awareness skills; Nonjudgment subscale score range: 8-40, higher scores = greater nonjudgment skills; Nonreactivity subscale score range: 7-35, higher scores = greater nonreactivity skills
State Mindfulness | Weeks 1, 3, 6
  State Mindfulness Scale for Physical Activity; 2 subscales, each with score range: 0-24, higher scores = higher levels of mindfulness
Interoceptive Awareness | Week 0, week 3, post-intervention (after 6 week intervention)
  Multidimensional Assessment of Interoceptive Awareness; 8 subscales, each with score ranges: 0-5, higher scores = better

CONTACTS AND LOCATIONS:
Locations (1):
- BIDMC, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No